CLINICAL TRIAL: NCT04157231
Title: Essential Acute Stroke Care in Low Resource Settings: a Pilot Study
Acronym: EASY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: World Heart Federation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: GI_NM-01-2019
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Acute Stroke
Keywords: Stroke; Ischemic stroke; hemorrhagic stroke; stroke package
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Intervention Model Description: A before and after, effectiveness-implementation hybrid study design with blinded outcome assessment will be conducted. This type 1 effectiveness-implementation hybrid design will test the essential acute stroke care management plan and secondarily gather data to inform subsequent research trials
Who Masked: Outcomes Assessor
Masking Description: The clinical outcome will be assessed by a blinded assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care to be provided to patients as per hospital guidelines for 3 months
- Intervention arm (Other): The intervention consists of training and education of the site staff about the treatment protocol for the different components of the management plan will be provided on two occasions. This intervention will run for 3 months.
  Refresher training will be given monthly during the intervention.
  Interventions: Other: Acute stroke care Intervention arm

INTERVENTIONS:
Other: Acute stroke care Intervention arm — Training and education of the site staff about the treatment protocol for the different components of the management plan will be provided on two occasions. The aim of these sessions will be to educate stroke champions and other site staff on the management protocols. Available training resources will be accessed (including online materials) and simulation training will be used. New skills such as dysphagia assessment will be emphasized based on existing knowledge and competencies. After training, staff will have another assessment (Post-test) in order to determine whether they have been adequately trained and are able to adhere to the essential acute stroke care management plan. A standardised Power Point presentation and accompanying handouts will be made available for further use in the ward.
  Refresher training will be provided monthly during the intervention.
  Arms: Intervention arm

SUMMARY:
An investigator-initiated, evaluator-blinded, prospective, multi centre, before-and-after, effectiveness-implementation hybrid design study to assess the feasibility of essential acute stroke care in a low resource setting

DETAILED DESCRIPTION:
This is a multicentre, before and after, effectiveness-implementation hybrid study design with blinded outcome assessment. Patients admitted to the participating hospitals will be managed under usual care conditions for three months (control arm). This will be followed by the training of the doctors and nurses in those hospitals on essential acute stroke care management. Patient management for the following three months after the training (intervention) will then be assessed to evaluate its impact on the care and clinical outcome of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years)
* A clinical or imaging-based diagnosis of acute stroke (ischemic or haemorrhagic) within 72 hours of stroke symptom onset
* Provision of written informed consent
* Subjects in observational, natural history and/or epidemiological studies not involving an intervention are eligible.

Exclusion Criteria:

* Patients who have undergone intravenous thrombolysis or mechanical thrombectomy
* Patients who are planned for transfer to the intensive care unit
* Subarachnoid haemorrhage
* Participation in an interventional medical investigation or clinical trial currently or within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Adherence | 30 days
  Primary Outcome Measure: Adherence to the predefined components of the essential acute stroke care management plan Adherence will be expressed as all or none measure and is defined as the proportion of patients who receive all the components of acute stroke care management for which the patient is eligible. Adherence will also be expressed as a composite measure, which is defined as the total number of eligible components performed divided by the total number of components for which the patient was eligible.

SECONDARY OUTCOMES:
Death or disability | 30 Days
  Death or disability as measured by Modified Rankin Scale (mRS) at 30 days. The mRS is a disability scale that ranges from 0 (no symptoms) to 6 (death).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Abanto, Dr, Principal Investigator — National Institute of Neurological Sciences, Lima, Peru; Kolawawole Wahab, Professor, Principal Investigator — University of Ilorin & University of Ilorin Teaching Hospital Ilorin, Nigeria; Hasan Farhan, Professor, Principal Investigator — President of Iraqi Scientific Council of Cardiology,Iraq; Yi Sui, Dr, Principal Investigator — Shenyang First People's Hospital Hospital Affiliated Brain Hospital; Saima Hilal, A/Professor, Principal Investigator — National University of Singapore; Lily Song, Dr, Principal Investigator — The George Institute of Global Health, China; Craig Anderson, Professor, Principal Investigator — Executive Director The George Institute for Global Health - China
Locations (4):
- Nigeria (2):
  - Murtala Muhammad Specialist Hospital, Kano, Kano State
  - Federal Medical Centre, Lokoja, Kogi State
- Peru (2):
  - Hospital de Apoyo II-2 Sullana, Piura
  - Hospital de la Amistad Peru Corea Santa Rosa II-2, Piura

IPD SHARING:
Plan to Share IPD: Yes
Requests for access to the de-identified data that underlie the study results should be made to: datasharing@georgeinstitute.org.
  We will provide data to researchers with a methodologically sound proposal, and will work with interested parties to define and operationalise a data access agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after publication of the main paper